CLINICAL TRIAL: NCT03574402
Title: An Open-label, Multi-center, Phase II Umbrella Study to Assess Efficacy of Targeted Therapy or Immunotherapy Directed by Next Generation Sequencing (NGS) in Chinese Patients With Advanced NSCLC (TRUMP)
Brief Title: Phase II Umbrella Study Directed by Next Generation Sequencing
Acronym: TRUMP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Collaborators: Chinese Thoracic Oncology Group (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG1702
Record Dates: First submitted 2018-06-20; First posted 2018-07-02 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC; advanced stage; high throughput sequencing; targeted therapy; immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — abivertinib; Afatinib; Crizotinib; ensartinib; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; AZD3759; nimotuzumab; Pemetrexed; Cisplatin; sintilimab; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (18):
- Arm1: Avitinib Maleate (Experimental): Patients with EGFR de novo T790m mutation receive Avitinib 300mg orally (PO) twice daily (BID) on day 1-28.
  Interventions: Drug: Avitinib Maleate
- Arm2: Chidamide plus Afatinib (Experimental): Patients with EGFR sensitive mutation with BIM deletion polymorphism receive Afatinib plus Chidamide.
  Chidamide will be administered 30mg orally twice weekly, 28 days as one cycle. Afatinib will be administered 40mg orally once a day, 28 days as one cycle.
  Interventions: Drug: Afatinib; Drug: Chidamide
- Arm3: crizotinib (Experimental): Patients with MET 14 exon mutation receive crizotinib 250mg PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Crizotinib
- Arm4: X396 (Experimental): Patients with MET amplification receive X396 225mg PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: X-396
- Arm5: X396 (Experimental): Patients with ROS1 fusion receive X396 225mg PO QD on days 1-28. 28 days as one cycle. Courses repeat every 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: X-396
- Arm6: X396 (Experimental): Patients with Ntrk1/2/3 fusion receive X396 225mg PO QD on days 1-28. 28 days as one cycle. Courses repeat every 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: X-396
- Arm7: Pyrotinib Maleate (Experimental): Patients with HER2 mutation receive Pyrotinib Maleate 400mg PO QD on days 1-28. 28 days as one cycle. Courses repeat every 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pyrotinib Maleate
- Arm8: AZD3759 (Experimental): EGFR sensitive mutation with brain/meningeal metastasis receive AZD3759 200mg PO BID on days 1-28. 28 days as one cycle. Courses repeat every 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: AZD3759
- Arm9: Pirotinib (Experimental): Patients with EGFR20ins mutation positive receive Pirotinib.
  This arm was divided into three groups:
  Group 1, 60mg PO QD on days 1-28. 28 days as one cycle. Group 2, 40mg PO BID on days 1-28. 28 days as one cycle. Group 3, Dosage was determined according to the number of PR patients in Group 2.
  Interventions: Drug: Pirotinib
- Arm10: Nimotuzumab plus gemcitabine and carboplatin (Experimental): Lung squamous cell carcinoma with EGFR amplification. Nimotuzumab 400mg, iv gtt. on day 1,8,15. Gemcitabine 1250mg/m^2, iv gtt. on day 1,8. Carboplatin AUC5, iv gtt. Q3W on day 1.
  21 days as one cycle. Courses repeat every 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Nimotuzumab; Drug: Gemcitabine; Drug: Carboplatin
- Arm11: Nimotuzumab plus pemetrexed and cisplatin (Experimental): Lung adenocarcinoma with EGFR amplification. Nimotuzumab 400mg, iv gtt. on day 1,8,15. pemetrexed 500mg/m^2, iv gtt. on day 1. Cisplatin 75mg/m^2, iv gtt. Q3W on day 1.
  21 days as one cycle. Courses repeat every 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Nimotuzumab; Drug: Pemetrexed; Drug: Cisplatin
- Arm12: Pirotinib (Experimental): Patients with rare EGFR mutation receive Pirotinib.
  This arm was divided into two groups:
  Group 1, 40mg PO BID on days 1-28. 28 days as one cycle. Group 2, Dosage was determined according to the number of PR patients in Group 1.
  Interventions: Drug: Pirotinib
- Arm13: Avitinib (Experimental): Patients with EGFR sensitive mutation receive Avitinib 300mg PO BID on days 1-28. 28 days as one cycle. Courses repeat every 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avitinib Maleate
- Arm14: Sintilimab (Experimental): Patients with PD-L1(TPS)≥50% without EGFR mutation or ALK rearrangement. Sintilimab 200mg iv gtt. Q3W on day1. 21 days as one cycle. Courses repeat every 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Sintilimab
- Arm15: Sintilimab (Experimental): Patients with TMB≥10 mut/Mb，1%≦PD-L1<50% without EGFR mutation or ALK rearrangement.
  Sintilimab 200mg iv gtt. Q3W on day1. 21 days as one cycle. Courses repeat every 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Sintilimab
- Arm16: Sintilimab (Experimental): Patients with KRAS and TP53 mutation, 1%≦PD-L1<50%, TMB<10 mut/Mb without EGFR mutation or ALK rearrangement.
  Sintilimab 200mg iv gtt. Q3W on day1. 21 days as one cycle. Courses repeat every 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Sintilimab
- Arm17: Sintilimab plus pemetrexed and cisplatin (Experimental): Patients with PD-L1<1%, TMB<10 mut/mb without EGFR mutation, ALK rearrangement, KRAS or TP53 mutation.
  Sintilimab 200mg iv gtt. Q3W on day1. Pemetrexedb 500mg/m^2 iv gtt. Q3W on day1. Cisplatin 75mg/m^2 iv gtt. Q3W on day1. 21 days as one cycle. Courses repeat every 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Sintilimab
- Arm18: Sintilimab plus Gemcitabine and carboplatin (Experimental): Patients with PD-L1<1%, TMB<10 mut/mb without EGFR mutation, ALK rearrangement, KRAS or TP53 mutation.
  Sintilimab 200mg iv gtt. Q3W on day1. Gemcitabine 1g/m^2 iv gtt. on day1,8. Carboplatin AUC5 iv gtt. Q3W on day1. 21 days as one cycle. Courses repeat every 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Sintilimab; Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Avitinib Maleate — 300mg orally (PO) twice daily (BID) on day 1-28.
  Other Names: AC0010
  Arms: Arm13: Avitinib; Arm1: Avitinib Maleate
Drug: Afatinib — 40mg orally once a day, 28 days as one cycle.
  Other Names: Giotrif
  Arms: Arm2: Chidamide plus Afatinib
Drug: Crizotinib — 250mg PO QD on days 1-28. 28 days as one cycle.
  Other Names: Xalkori
  Arms: Arm3: crizotinib
Drug: X-396 — 225mg PO QD on days 1-28. 28 days as one cycle.
  Other Names: ensartinib
  Arms: Arm4: X396; Arm5: X396; Arm6: X396
Drug: Chidamide — 30mg orally twice weekly, 28 days as one cycle.
  Other Names: Epidaza
  Arms: Arm2: Chidamide plus Afatinib
Drug: Pyrotinib Maleate — 400mg PO QD on days 1-28. 28 days as one cycle.
  Other Names: SHR1258
  Arms: Arm7: Pyrotinib Maleate
Drug: AZD3759 — 200mg PO BID on days 1-28. 28 days as one cycle.
  Arms: Arm8: AZD3759
Drug: Pirotinib — 60mg PO QD/40mg PO BID on days 1-28. 28 days as one cycle.
  Other Names: KBP-5209
  Arms: Arm12: Pirotinib; Arm9: Pirotinib
Drug: Nimotuzumab — 400mg, iv gtt. on day 1,8,15. 21 days as one cycle.
  Arms: Arm10: Nimotuzumab plus gemcitabine and carboplatin; Arm11: Nimotuzumab plus pemetrexed and cisplatin
Drug: Pemetrexed — 500mg/m^2, iv gtt. Q3W. 21 days as one cycle.
  Other Names: LY231514
  Arms: Arm11: Nimotuzumab plus pemetrexed and cisplatin; Arm17: Sintilimab plus pemetrexed and cisplatin
Drug: Cisplatin — 75mg/m^2, iv gtt. Q3W on day1. 21 days as one cycle.
  Other Names: CDDP
  Arms: Arm11: Nimotuzumab plus pemetrexed and cisplatin; Arm17: Sintilimab plus pemetrexed and cisplatin
Drug: Sintilimab — 200mg iv gtt. Q3W on day1. 21 days as one cycle.
  Arms: Arm14: Sintilimab; Arm15: Sintilimab; Arm16: Sintilimab; Arm17: Sintilimab plus pemetrexed and cisplatin; Arm18: Sintilimab plus Gemcitabine and carboplatin
Drug: Gemcitabine — 1g/m^2 iv gtt. on day1,8. 21 days as one cycle.
  Other Names: LY188011
  Arms: Arm18: Sintilimab plus Gemcitabine and carboplatin
Drug: Gemcitabine — 1.25g/m^2 iv gtt. on day1,8. 21 days as one cycle.
  Other Names: LY188011
  Arms: Arm10: Nimotuzumab plus gemcitabine and carboplatin
Drug: Carboplatin — AUC5 iv gtt. Q3W on day1. 21 days as one cycle.
  Other Names: NSC 241240
  Arms: Arm10: Nimotuzumab plus gemcitabine and carboplatin; Arm18: Sintilimab plus Gemcitabine and carboplatin

SUMMARY:
This phase II, umbrella trial study directed by next generation sequencing (NGS) works in Chinese patients with advanced stage NSCLC who never received any anti-tumor treatment. The purpose of this study is to evaluate efficacy of targeted therapies or immunotherapy to NSCLC patients whose tumor harbors a genomic variant known to be a drug target or to predict sensitivity to a drug.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the anti-tumor efficacy of targeted agents or checkpiont inhibitors in advanced stage NSCLC with genomic alteration.

SECONDARY OBJECTIVES:

I. To evaluate the clinical efficacy of targeted agents or checkpiont inhibitors in advanced stage NSCLC with genomic alteration.

II. To evaluate safty and tolerence of targeted agents or checkpiont inhibitors in advanced stage NSCLC with genomic alteration.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed, unresectable stage IIIB or stage IV NSCLC
2. Patients who have never received any anticancer treatment regimen Note: Patients that have received adjuvant or neoadjuvant chemotherapy and developed metastatic disease after 12 months from the end of that therapy would be eligible for enrollment.
3. Measurable disease according to RECIST v.1.1 (Irradiated lesions are not considered measurable unless they have clearly progressed since radiotherapy)
4. With or without brain or leptomeningeal metastasis (BM/LM). For patients with symptoms of BM/LM, no need for local therapy should be confirmed by investigator and no dramatic decline of performance status in 2 weeks.
5. ECOG performance status ≤ 2
6. Expected survival > 12 weeks
7. Patients must be suitable and willing to undergo mandatory tumor biopsy according to treating institution's guidelines and requirements for such procedure if there is no archival biopsy available.
8. Provision of signed and dated written informed consent by the patient or legally acceptable representative prior to any study-specific procedures.
9. Palliative radiotherapy was allowed before enrollment, and radiotherapy-related toxicity grade should no more than 1 (ctcae4.03).
10. No anti-tumor Chinese medicine has been used in the past, or has been used for no more than 3 doses, and stopped for more than 2 weeks before enrollment.
11. Absolute neutrophil count (ANC) ≥ 1.5x10^9/L without the use of growth factor in the past 14 days. Platelets ≥ 90 × 10^9/L without blood transfusion in the past 14 days. Hemoglobin > 9g/dL.
12. Negative pregnancy test (only for women with pregnancy possibility). No possibility of pregnancy defined as at least one year after menopause, or having undergone surgical sterilization or hysterectomy. All patients (male or female) agreed to take contraceptive measures during the treatment and within 8 weeks after the treatment.

Exclusion Criteria:

1. Active hepatitis (HBsAg positive and HBV copy number in upper limit of normal)
2. Previous or current active interstitial lung disease (ILD)
3. Patients known to be HIV positive or with other acquired, congenital immunodeficiency diseases, or with a medical history of organ transplantation.
4. Major surgery ≤ 2 weeks prior to study entry.
5. Any other malignancies within the last 5 years before study enrollment, except for un completely resected basal cell carcinoma, in situ bladder cancer, cervical carcinoma in situ.
6. Patients previously treated with the investigational drugs or known to be allergic to ingredients or excipients of the investigational drugs.
7. Pregnant or lactating women.
8. Patients with swallowing dysfunction, active gastrointestinal disease or other diseases that significantly affect the absorption, distribution, metabolism and excretion of oral drugs. The patients who have had subtotal gastrectomy before. (this standard is applicable to the arms with oral drugs only)
9. Body temperature above 38 ℃ in the past week, or there was active infection with clinical significance. Active tuberculosis;
10. Evidence of serious or uncontrollable systemic diseases (such as severe mental, neurological, epilepsy or dementia, unstable or uncompensated respiratory, cardiovascular, liver or kidney diseases, uncontrolled hypertension [higher than CTCAE Level 3 hypertension after drug treatment]);
11. Patients with bleeding tendency or taking anticoagulants ;
12. There are significant clinical abnormalities in rhythm, conduction or morphology of resting ECG, such as complete left bundle branch block, heart block above degree II, clinically significant ventricular arrhythmia or atrial fibrillation, unstable angina, congestive heart failure, chronic heart failure with NYHA grade ≥ 2.
13. Myocardial infarction, coronary / peripheral artery bypass or cerebrovascular accident occurred within 3 months.
14. QTc of 12 lead ECG was ≥ 450 ms in male and ≥ 470 ms in female;
15. Diagnosed with another malignant disease in the past five years besides NSCLC.
16. More than 30% of the bone marrow had received radiotherapy within 4 weeks before treatment.
17. Any drugs known to extend QT interval were being used within 2 weeks prior to first administration.
18. Strong CYP3A4 inhibitor/inductionor or CYP3A4 substrate were used within 2 weeks, including but not limited to azanavir, clarithromycin, inddenavir, itraconazole, ketoconazole, nefazodone, nefinavir, ritonavir, xaquinavir, talicamycin, acesodamycin, voriconazole, carbamazepine, phenobarbital, phenytoin, rifampin, rifampin, Hypericum perforatum, dihydroergotamine, ergotamine, pimozite, astemizole, cisapride and terfenadine.
19. Strong P-gp inhibitor was used within 2 weeks (including but not limited to verapamil, cyclosporine A and right verapamil).
20. Other potential risks that are not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Response rate (RR) | 24 months
  RECIST version 1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 24 months
  RECIST version 1.1
Overall survival (OS) | 48 months
  Overall Survival is defined as the time from first dose to death due to any cause. Through the follow-up within 30 days after study completion or termination of the last subject, death and date of death will be checked for subject alive during treatment period
Disease control rate（DCR） | 24 months
  RECIST version 1.1
Duration of response (DOR) | 24 months
  RECIST version 1.1
Toxicity (number of patients with treatment-related AE as assessed by CTCAE v4.03) | 24 months
  number of patients with treatment-related AE as assessed by CTCAE v4.03
Health-Related Quality of Life (HRQOL) | 24 months
  EORTC-LC13
To explore the mechanism of drug resistance in the treatment of specific gene mutation | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Long Wu, Study Chair — Guangdong Association of Clinical Trials
Locations (1):
- Guangdong Lung Cancer Institute, Guangdong Provincial People's Hospital, Guangdong Academy of Medical Sciences, School of Medicine, South China University of Technology, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Liu SM, Tu HY, Wei XW, Yan HH, Dong XR, Cui JW, Zhou Z, Xu CR, Zheng MY, Li YS, Wang Z, Bai XY, Li AN, Sun YL, Huang J, Lin JX, Ke EE, Xu BF, Lu C, Du Y, Chen Y, Ma R, Wang BH, Cang SD, Wang BC, Chen HJ, Yang JJ, Li Y, Zhou Q, Wu YL. First-line pyrotinib in advanced HER2-mutant non-small-cell lung cancer: a patient-centric phase 2 trial. Nat Med. 2023 Aug;29(8):2079-2086. doi: 10.1038/s41591-023-02461-x. Epub 2023 Jul 24. PMID 37488286
- [Derived] Liu SM, Yan HH, Wei XW, Lu C, Dong XR, Du Y, Cui JW, Chen Y, Ma R, Wang BH, Zhou Z, Cang SD, Yang JJ, Tu HY, Zhang XC, Zhong WZ, Zhou Q, Wu YL. Biomarker-Driven Studies With Multi-targets and Multi-drugs by Next-Generation Sequencing for Patients With Non-Small-Cell Lung Cancer: An Open-Label, Multi-center, Phase II Adaptive Umbrella Trial and a Real-World Observational Study (CTONG1702&CTONG1705). Clin Lung Cancer. 2022 Nov;23(7):e395-e399. doi: 10.1016/j.cllc.2022.05.009. Epub 2022 May 11. PMID 35659479